CLINICAL TRIAL: NCT01106430
Title: A Phase 3b, Double-blind, Randomised, Active-controlled, Parallel Group Study to Assess the Time to Response of Lisdexamfetamine Dimesylate to Atomoxetine Hydrochloride in Children and Adolescents Aged 6-17 Years With Attention-Deficit/Hyperactivity Disorder (ADHD) Who Have Had an Inadequate Response to Methylphenidate Therapy
Brief Title: Comparison of Lisdexamfetamine Dimesylate With Atomoxetine HCl in Attention-Deficit/Hyperactivity Disorder (ADHD) Subjects With an Inadequate Response to Methylphenidate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD489-317; 2009-011745-94 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-19 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine Dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Atomoxetine Hydrochloride (Active Comparator)
  Interventions: Drug: Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Oral 30, 50, or 70mg once-daily for 9 weeks
  Other Names: Vyvanse
  Arms: Lisdexamfetamine Dimesylate
Drug: Atomoxetine Hydrochloride — Oral 10mg to 100mg once-daily for 9 weeks
  Other Names: Strattera
  Arms: Atomoxetine Hydrochloride

SUMMARY:
This study will evaluate how long it takes for ADHD symptoms to improve in subjects who are judged by the Investigator to have had an inadequate response to methylphenidate therapy. The study will also test the safety of Lisdexamfetamine Dimesylate and how well it works.

ELIGIBILITY:
Inclusion Criteria:

* Subject has had an historical or current inadequate response to methylphenidate (MPH) treatment. Inadequate response includes but is not limited to the presence of some residual symptoms, with associated impairment inadequate duration of action and/or variability of symptom control, and/or Investigator feels that the subject may derive benefit from an alternative drug treatment to MPH therapy.
* Subject is a male or female aged 6-17 years inclusive at the time of consent
* Subject must meet Diagnostic and Statistical Manual of Mental Disorders, fourth edition. - Text Revision (DSM IV TR) criteria for a primary diagnosis of ADHD based on a detailed psychiatric evaluation
* Subject must have a baseline ADHD-RS-IV total score 28.

Exclusion Criteria:

* Subject has taken more than 1 MPH treatment (for example, 2 or more different MPH treatments). Examples include but are not limited to RITALIN immediate release (IR) and EQUASYM IR; MEDIKINET IR and CONCERTA; RITALIN long-acting LA and CONCERTA. Note: this does not include subjects who have taken IR MPH for dose titration on a short-term basis (for example, £4 weeks) with an adequate response
* In the Investigator's judgement, subject has failed to respond to more than 1 previous course(s) of MPH treatment. Failure to respond includes worsening of symptoms or no change/minimal improvement of symptoms.
* Subject has previously been exposed to STRATTERA or to amphetamine therapy
* Subject has previously demonstrated intolerable side effects to 1 MPH treatment which limited titration to acceptable efficacy or that required a decrease in dose resulting in unacceptable tolerability and/or efficacy
* Subject has a current, controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as any severe comorbid Axis II disorder or severe Axis I disorder or other symptomatic manifestations, such as agitated states, marked anxiety, or tension that, in the opinion of the examining physician, will contraindicate treatment with SPD489 or STRATTERA or confound efficacy or safety assessments.
* Subject has a conduct disorder. Oppositional Defiant Disorder is not exclusionary.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2010-06-28 (Actual); Primary Completion 2012-07-19 (Actual); Study Completion 2012-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (64):
- United States (34):
  - Harmonex Neuroscience Research, Inc, Dothan, Alabama
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Shanti Clinical Trials, Colton, California
  - Psychiatric Centers at San Diego Feighner Research, San Diego, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Fidelity Clinical Research, Inc., Lauderhill, Florida
  - Clinical Neuroscience Solutions, INC, Orlando, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Psychiatric Associates, Naperville, Illinois
  - Clinco, Terre Haute, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Four Rivers Clinical Research, Inc, Paducah, Kentucky
  - Louisianna Research Associates, New Orleans, Louisiana
  - Office of Marc Hertzman, MD, PC, Rockville, Maryland
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Midwest Research Group/Saint Charles Psychiatric Associates, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Children's Specialized Hospital, Toms River, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Triangle Neuropsychiatry, PLLC, Durham, North Carolina
  - Innovis Health, Fargo, North Dakota
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - CRI Worldwide, LLC Kirkbride Division, Philadelphia, Pennsylvania
  - Future Search Clinical Trials, Austin, Texas
  - Red Oak Psychiatry Association, PA, Houston, Texas
  - Western Clinical Investigations, Lubbock, Texas
  - Cerebral Research, LLC, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Eastside Therapeutic Resource, Kirkland, Washington
- Belgium (2):
  - ZiekenhuisNetwerk Antwerpen, Hoboken, Antwerpen
  - Universitair Ziekenhuis Gasthuisberg, Leuven, Flemish Brabant
- Canada (5):
  - Child and Adolescent Centre, Edmonton, Alberta
  - Centre for Anxiety Attention Deficit and Trauma, Hamilton, Ontario
  - AK Karan Holdings, Ltd., Oakville, Ontario
  - The Kids Clinic, Whitby, Ontario
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Germany (6):
  - Albert-Ludwigs-Universitat Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Zentralinstitut für Seelische Gesundheit Mannheim, Mannheim, Baden-Wurttemberg
  - Schwerpunktpraxis für Entwicklung und Lernen, Bamberg, Bavaria
  - Medizinisches Studienzentrum Würzburg, Würzburg, Bavaria
  - Klinikum Frankfurt/Oder, Frankfurt (Oder), Brandenburg
  - Praxis Dr. Wolff, Hagen, North Rhine-Westphalia
- Hungary (4):
  - Szegedi Tudományegyetem Gyermek es lfjusagpszichlatrlai Osztaly, Szeged, Csongrád megye
  - Vadaskert Korhaz es Szakambulancia Gyermek es lfjusagpszichiatria, Budapest
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Gyermek- es lfjusagpszichiatriai Szakrendeles es Gondozo, Pécs
- Azienda Ospedaliero-Universitaria di Cagliari, Cagliari, Italy
- Poland (2):
  - Katedra i Klinika Psychiatarii, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw, Masovian Voivodeship
- Spain (6):
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Marítimo, Unidad de Salud Mental Infanto-Juvenil (USMI-J, Torremolinos, Malaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Complejo Hospitalario Universitario de Badajoz, Badajoz
  - Hospital Clinic i Provincial de Barcelona, Barcelona
- Sweden (2):
  - Drottning Silvias Barnsjukhus, Gothenburg
  - Astrid Lindgren Children's Hospital/Karolinska University Hospital, Stockholm
- United Kingdom (2):
  - Basildon Hospital, Basildon, Essex
  - Tayside Children's Hospital, Dundee, Scotland

REFERENCES:
- [Result] Dittmann RW, Cardo E, Nagy P, Anderson CS, Bloomfield R, Caballero B, Higgins N, Hodgkins P, Lyne A, Civil R, Coghill D. Efficacy and safety of lisdexamfetamine dimesylate and atomoxetine in the treatment of attention-deficit/hyperactivity disorder: a head-to-head, randomized, double-blind, phase IIIb study. CNS Drugs. 2013 Dec;27(12):1081-92. doi: 10.1007/s40263-013-0104-8. PMID 23959815
- [Derived] Nagy P, Hage A, Coghill DR, Caballero B, Adeyi B, Anderson CS, Sikirica V, Cardo E. Functional outcomes from a head-to-head, randomized, double-blind trial of lisdexamfetamine dimesylate and atomoxetine in children and adolescents with attention-deficit/hyperactivity disorder and an inadequate response to methylphenidate. Eur Child Adolesc Psychiatry. 2016 Feb;25(2):141-9. doi: 10.1007/s00787-015-0718-0. Epub 2015 May 22. PMID 25999292
- [Derived] Dittmann RW, Cardo E, Nagy P, Anderson CS, Adeyi B, Caballero B, Hodgkins P, Civil R, Coghill DR. Treatment response and remission in a double-blind, randomized, head-to-head study of lisdexamfetamine dimesylate and atomoxetine in children and adolescents with attention-deficit hyperactivity disorder. CNS Drugs. 2014 Nov;28(11):1059-69. doi: 10.1007/s40263-014-0188-9. PMID 25038977

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisdexamfetamine Dimesylate: Lisdexamfetamine Dimesylate (LDX, Vyvanse, SPD489) was administered orally once-daily at approximately 7:00am for 9 weeks (4-week dose optimization period and a 5-week dose maintenance period) at doses of either 30, 50, or 70 mg.
- Atomoxetine Hydrochloride: Atomoxetine Hydrochloride (Strattera) was administered orally once-daily at approximately 7:00am for 9 weeks (4-week dose optimization period and a 5-week dose maintenance period) at weight adjusted doses of 10 mg to 100 mg.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Started | 133 | 134
Completed | 100 | 101
Not Completed | 33 | 33
Not completed — Adverse Event | 8 | 10
Not completed — Lack of Efficacy | 2 | 13
Not completed — Lost to Follow-up | 5 | 1
Not completed — Early Termination Requested By Sponsor | 1 | 0
Not completed — Moved Out Of State | 0 | 1
Not completed — Refused To Take Medication | 0 | 1
Not completed — Noncompliance | 0 | 1
Not completed — Hard Time Swallowing The Pills | 1 | 0
Not completed — Previous Use Of Marijuana | 1 | 0
Not completed — Protocol Violation | 7 | 2
Not completed — Withdrawal by Subject | 8 | 4

BASELINE CHARACTERISTICS:
Population: Safety Population was used for baseline characteristics (n = 262). Defined as all subjects who were randomized and who had taken at least 1 dose of investigational product. Five randomized subjects did not take any investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride | Total
Number analyzed (Participants) | 128 | 134 | 262
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.9 (3.01) | 10.4 (2.84) | 10.6 (2.93)
Age, Customized [Count of Participants; unit: Participants]
  13 - 17 years | 34 | 34 | 68
  6 - 12 years | 94 | 100 | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 31 | 65
  Male | 94 | 103 | 197
Region of Enrollment [Count of Participants; unit: Participants] — All enrolled subjects defined as all randomized subjects (n = 267).
  Participants
    BELGIUM | 0 | 2 | 2
    CANADA | 17 | 18 | 35
    GERMANY | 20 | 22 | 42
    HUNGARY | 10 | 10 | 20
    ITALY | 1 | 0 | 1
    POLAND | 0 | 1 | 1
    SPAIN | 12 | 10 | 22
    SWEDEN | 3 | 3 | 6
    UNITED STATES | 70 | 68 | 138

OUTCOME MEASURES:

1. Primary Outcome: Time to First Response
Description: Time to first response was defined as a Clinical Global Impression-Improvement (CGI-I) value of 1 (very much improved) or 2 (much improved) first recorded following first dose of investigational product. CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Time Frame: 9 weeks
Population: Full Analysis Set defined as all subjects who were randomized and who had taken at least 1 dose of investigational product. One subject was randomized to receive Strattera, but actually received Lisdexamfetamine Dimesylate. For all efficacy analyses this subject is included in the Strattera arm per the intention to treat principle.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 127 | 135
Days | 12.0 [8.0 to 16.0] | 21.0 [15.0 to 23.0]
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.001, Peto-Peto-Prentice Wilcoxon Test

2. Secondary Outcome: Percent of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores - Last Observation Carried Forward (LOCF)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 9 weeks
Population: Full Analysis Set defined as all subjects who were randomized and who had taken at least 1 dose of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 126 | 132
percentage of participants | 81.7 | 63.6
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 18.1, 95% CI 2-sided [7.5 to 28.7]

3. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-Fourth Edition (ADHD-RS-IV) Total Score at 9 Weeks - LOCF
Description: ADHD-RS-IV consists of 18 items scored on a 4-point scale from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. A decrease in score indicates an improvement in ADHD symptomology.
Time Frame: Baseline and 9 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 126 | 133
units on a scale | -26.1 (1.16) | -19.7 (1.13)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in LS Means = -6.5, 95% CI 2-sided [-9.3 to -3.6]

4. Secondary Outcome: Change From Baseline in the Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Global Score at Up to 9 Weeks
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and up to 9 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 107 | 113
units on a scale | -0.35 (0.034) | -0.27 (0.032)
Statistical Analysis 1: Comparison: Lisdexamfetamine Dimesylate vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.046, ANCOVA; Difference in LS Means = -0.09, 95% CI 2-sided [-0.17 to -0.00]

5. Secondary Outcome: Health Utilities Index-2 (HUI-2) Scores at Up to 9 Weeks
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status.
Time Frame: up to 9 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 116 | 123
units on a scale | 0.920 (0.0961) | 0.922 (0.0937)

6. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale for Children (BPRS-C) Total Score at Up to 9 Weeks
Description: The BPRS-C characterizes psychopathology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology.
Time Frame: Baseline and up to 9 weeks
Population: Safety Population defined as all subjects who were randomized and who had taken at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 117 | 123
units on a scale | -10.7 (9.27) | -7.9 (9.07)

7. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: 9 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 127 | 132
participants
  Suicidal ideation | 0 | 0
  Suicidal behavior | 0 | 0

8. Secondary Outcome: Udvalg for Kliniske Undersogelser Side Effect Rating Scale - Clinician (UKU-SERS-Clin) With Side Effects Scores >=1
Description: UKU-SERS-Clin is composed of 48 items each of which asks about a single side effect. Each side effect is rated based on a 4-point scale ranging from 0 (no or doubtful presence) to 3 (the least favorable rating). The rating is independent of whether the symptom is regarded as related to the investigational product.
Time Frame: 9 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Number analyzed (Participants) | 127 | 132
participants
  Weight Loss | 46 | 19
  Reduced Duration of Sleep | 29 | 16
  Asthenia/Lassitude/Increased Fatigability | 25 | 29
  Tension/Inner Unrest | 20 | 22
  Nausea/Vomiting | 19 | 26
  Sleepiness/Sedation | 16 | 35
  Reduced Salivation | 16 | 6
  Headache-Tension Headache | 15 | 17
  Concentration Difficulties | 75 | 92
  Failing Memory | 10 | 21
  Depression | 6 | 10
  Increased Duration of Sleep | 12 | 12
  Increased Dream Activity | 3 | 8
  Emotional Indifference | 12 | 10
  Dystonia | 0 | 1
  Rigidity | 0 | 1
  Hypokinesia/Akinesia | 1 | 0
  Hyperkinesia Logic | 2 | 3
  Tremor | 3 | 1
  Akathisia | 0 | 2
  Paraesthesias | 1 | 0
  Accomodation Disturbances | 0 | 2
  Increased Salivation | 1 | 2
  Diarrhea | 6 | 9
  Constipation | 9 | 5
  Micturition Disturbances | 0 | 1
  Polyuria/Polydipsia | 3 | 2
  Orthostatic Dizziness | 10 | 9
  Palpitations/Tachycardia | 1 | 5
  Increased Tendency to Sweating | 3 | 5
  Rash-Morbiliform | 0 | 1
  Rash-Petechial | 1 | 0
  Rash-Urticarial | 1 | 1
  Rash-Cannot be Classified | 1 | 2
  Pruritus | 4 | 7
  Weight Gain | 1 | 0
  Headache-Migraine | 2 | 2
  Headache-Other Forms | 11 | 10

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who were randomized and who had taken at least 1 dose of investigational product.
Arm/Group | Lisdexamfetamine Dimesylate | Atomoxetine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/134
Other Adverse Events (participants affected / at risk) | 92/128 | 95/134
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine Dimesylate (N=128) | Atomoxetine Hydrochloride (N=134)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 8 (10)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (3) | 10 (12)
CONSTIPATION (Gastrointestinal disorders) | 8 (9) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 9 (11)
DRY MOUTH (Gastrointestinal disorders) | 8 (8) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 16 (16) | 21 (27)
VOMITING (Gastrointestinal disorders) | 6 (6) | 13 (17)
FATIGUE (General disorders) | 12 (14) | 14 (16)
IRRITABILITY (General disorders) | 8 (8) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 8 (9) | 8 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 8 (8)
WEIGHT DECREASED (Investigations) | 28 (30) | 9 (9)
DECREASED APPETITE (Metabolism and nutrition disorders) | 33 (36) | 14 (14)
HEADACHE (Nervous system disorders) | 17 (25) | 22 (29)
SEDATION (Nervous system disorders) | 5 (5) | 8 (9)
SOMNOLENCE (Nervous system disorders) | 4 (4) | 16 (23)
INSOMNIA (Psychiatric disorders) | 15 (16) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.